CLINICAL TRIAL: NCT02223884
Title: A Study to Evaluate the Efficacy of Docetaxel and Carboplatin in Metastatic Malignant Melanoma Failed First-Line Dacabazine or Temozolomide Contained Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0300
Record Dates: First submitted 2014-08-17; First posted 2014-08-22 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Malignant Melanoma
Keywords: Malignant melanoma, second-line treatment, docetaxel, carboplatin
MeSH Terms: conditions — Melanoma | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- weekly docetaxel and carboplatin (Experimental)
  Interventions: Drug: docetaxel 35mg/m2; Drug: Carboplatin AUC3

INTERVENTIONS:
Drug: docetaxel 35mg/m2 — D1, 8 docetaxel 35 mg/m2 D1, 8 carboplatin AUC 3 every 3 weeks
Drug: Carboplatin AUC3 — D1, 8 docetaxel 35 mg/m2 D1, 8 carboplatin AUC 3 every 3 weeks

SUMMARY:
This is the phase II, single-arm, single-center study assessing the efficacy of weekly docetaxel plus carboplatin in second-line treatment of malignant melanoma (unresectable or metastatic) who has failed dacarbazine or temozolomide contained therapy. The primary end point is overall response rate according to RECIST 1.1 criteria assessed using CT or MRI and secondary end point includes disease control rate, progression free survival, overall survival and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven malignant melanoma (recurred or metastatic) that had progressed during or after receiving at least one cycle of a regimen containing dacarbazine or temozolomide in the advanced setting
* Measurable disease (RECIST)
* ECOG performance 0-2
* Adequate organ function
* Total bilirubin <1.5N ; ASAT and ALAT <2.5N
* Serum Creatinin < 1.5N
* ANC ≥ 1,500/mm³ (G-CSF allowed)
* Platelets ≥ 100,000/mm³
* Hb ≥ 9.0 g/dL
* Life expectancy of at least 12 weeks
* Signed Written Informed Consent

Exclusion Criteria:

* Symptomatic brain metastasis
* Previous history of treatment with taxane or platinum agent containing chemotherapy
* Previous major surgery within 2 weeks before the start of the trial, or a failure to recover from the surgery
* Previous history of other malignancies within 5 years except for cured skin basal cell carcinoma or cured in-situ cervix cancer
* Other severe medical conditions (infection, uncontrolled hypertension, heart failure, MI history within 6 months)
* Sensitivity to platinum agents or docetaxel
* Uncontrolled seizure
* Women pregnant or nursing
* Alcohol or drug abuser

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Response Rate | every 6 weeks, up to 4 year
  Response rate evaluation based on RECIST 1.1 confirmed by CT or MRI

SECONDARY OUTCOMES:
disease control rate | every 6 weeks, up to 4 year
progression free survival | every 6 weeks, up to 4 year
overall survival | every 6 weeks, up to 4 year
adverse events | every 6 weeks, up to 4 year

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea